CLINICAL TRIAL: NCT00295672
Title: Oral Vinorelbine and Cisplatin and Concurrent Radiotherapy After Induction Chemotherapy With Cisplatin-docetaxel in Patients With Locally Advanced Non-small-cell Lung Cancer. A Multicenter Phase II Trial
Brief Title: Oral Vinorelbine and Cisplatin and Concurrent Radiotherapy After Induction Chemotherapy in Locally Advanced NSCLC.
Acronym: VINCR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Fabre Clinic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB 05-110; VINCR - GFPC 05-03
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Lung Neoplasm
Keywords: Non-Small-Cell Lung,radiotherapy, Chemotherapy, vinorelbine
MeSH Terms: conditions — Lung Neoplasms | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vinorelbine

SUMMARY:
Our aim is to conducted a multicenter phase II trial of the cisplatin-oral vinorelbine -radiotherapy combination after induction chemotherapy with cisplatin-docetaxel in patient with NSCLC. Oral vinorelbine will be used in the present study rather than the intravenous form because: 1- Previous investigations have demonstrated that oral vinorelbine is as effective as the intravenous form in the treatment of NSCLC. 2 - We think that the use of oral agents in CT will reduce some disagreements provoked by intravenous injections: stress, infections, hemorrhage, displacement at the hospital and cost of CT.

.

DETAILED DESCRIPTION:
About one-third of patients with non-small-cell lung cancer (NSCLC) have inoperable, locally advanced stage III disease at diagnosis. The most satisfactory treatment for patients with locally advanced NSCLC is combination chemotherapy-radiotherapy (CT-RT). However, the optimal interval between irradiation and chemotherapy as well as the most effective chemotherapy protocol remains to be defined.

Our aim is to conducted a multicenter phase II trial of the cisplatin-oral vinorelbine -radiotherapy combination after induction chemotherapy with cisplatin-docetaxel in patient with NSCLC. Oral vinorelbine will be used in the present study rather than the intravenous form because: 1- Previous investigations have demonstrated that oral vinorelbine is as effective as the intravenous form in the treatment of NSCLC. 2 - We think that the use of oral agents in CT will reduce some disagreements provoked by intravenous injections: stress, infections, hemorrhage, displacement at the hospital and cost of CT.

Patients will be enrolled in the study by members of GFPC, a French cooperative group on thoracic oncology. The main eligibility criteria are : histologically or cytologically documented inoperable stage IIIA N2 or IIIB NSCLC previously untreated, absence of malignant pleural effusion, performance status (PS) =1 and patient life expectancy of at least 12 weeks. Induction chemotherapy will comprise two cycles of cisplatin 80mg/m2 and docetaxel 75mg/m2 (given on D1 and D22). Concomitant CT-RT will start on D57. Radiotherapy will occur from D57 until D99 (2 Gy/day, 5 days/week, total dose is 66 Gy). Cisplatin 80mg/m2 will be given on D57 (first day of irradiation) and D78. Oral vinorelbine 40 mg/m2 will be administered on D57, D64, D78 and D85. The main endpoint is the objective response rate. The tumor response will be assessed first at the end of induction chemotherapy, and again 4 weeks after concurrent CT-RT. Patients who will progress after induction chemotherapy will leave the study. Those with stable disease or a tumor response will receive the CT-RT combination. Tolerability, time until progression, duration of response and proportion of survival at 1, 2 and 3 years represent a secondary endpoints. The study will be achieved according to the French legislation and guidelines for biomedical research involving human subjects.

ELIGIBILITY:
Inclusion Criteria:

histologically or cytologically documented inoperable stage IIIA N2 or IIIB NSCLC previously untreated, absence of malignant pleural effusion, performance status (PS) =1 and patient life expectancy of at least 12 weeks.

Exclusion Criteria:

metastatic disease, small Cell lung carcinoma, prior chemotherapy, prior radiotherapy, resecable tumor, any instable systemic disease, any other malignancies within 5 years,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-02; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
TUMORAL RESPONSE (RECIST)
TOXICITY (NCI 20)

SECONDARY OUTCOMES:
SURVIVAL
TIME TO PROGRESSION
LATE RADIATION TOXICITY

CONTACTS AND LOCATIONS:
Overall Officials: gilles Robinet, Principal Investigator — CHU of Brest
Locations (6):
- France (6):
  - CHU of Brest, Brest
  - CH GAP, Gap
  - CHU de LIMOGES, Limoges
  - Hopital de la Croix Rousse, Lyon
  - Hôpital Sainte Margueritte, Marseille
  - CHU Hôpital Nord, Saint-Etienne

REFERENCES:
- [Background] Fournel P, Robinet G, Thomas P, Souquet PJ, Lena H, Vergnenegre A, Delhoume JY, Le Treut J, Silvani JA, Dansin E, Bozonnat MC, Daures JP, Mornex F, Perol M; Groupe Lyon-Saint-Etienne d'Oncologie Thoracique-Groupe Francais de Pneumo-Cancerologie. Randomized phase III trial of sequential chemoradiotherapy compared with concurrent chemoradiotherapy in locally advanced non-small-cell lung cancer: Groupe Lyon-Saint-Etienne d'Oncologie Thoracique-Groupe Francais de Pneumo-Cancerologie NPC 95-01 Study. J Clin Oncol. 2005 Sep 1;23(25):5910-7. doi: 10.1200/JCO.2005.03.070. Epub 2005 Aug 8. PMID 16087956
- [Background] Vergnenegre A, Daniel C, Lena H, Fournel P, Kleisbauer JP, Le Caer H, Letreut J, Paillotin D, Perol M, Bouchaert E, Preux PM, Robinet G; Groupe Francais de Pneumo-Cancerologie. Docetaxel and concurrent radiotherapy after two cycles of induction chemotherapy with cisplatin and vinorelbine in patients with locally advanced non-small-cell lung cancer. A phase II trial conducted by the Groupe Francais de Pneumo-Cancerologie (GFPC). Lung Cancer. 2005 Mar;47(3):395-404. doi: 10.1016/j.lungcan.2004.08.010. PMID 15713523
- See also: click here for more information — http://www.g-f-p-c.org